CLINICAL TRIAL: NCT02284269
Title: Meta-analysis in Post-Marketing Surveillances for Long-Term Drug Use of SGLT2 Inhibitors in Patients With Type 2 Diabetes Mellitus
Brief Title: Meta-analysis in Post-marketing Surveillances for SGLT2 Inhibitors in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pharmaceuticals and Medical Devices Agency, Japan (Other Government)
Responsible Party: Sponsor
Other Study IDs: PMDA-A2602
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SGLT2 Inhibitors — Ipragliflozin (Suglat®), Dapaglilozin (Forxiga®), Tofogliflozin (Deberza® / Apleway®), Luseogliflozin (Lusefi®), Canagliflozin (Canaglu®), Empagliflozin (Jardiance®)

SUMMARY:
The purpose of this study is to integrate the post-marketing surveillances data (Specified use-results surveys on long-term treatment) of the 6 SGLT2 inhibitors approved or applied in Japan and to evaluate the safety and efficacy of long-term use of each under actual clinical practice conditions.

In each post-marketing surveillance, 3000 patients who complete a 3 years treatment are enrolled. A total of 18000 patients are assessed in the meta-analysis.

ELIGIBILITY:
Patients with Type 2 diabetes mellitus starting medication of SGLT2 inhibitors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Type 2 diabetes mellitus starting medication of SGLT2 inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 3 years

SECONDARY OUTCOMES:
Incidence of cardiovascular events | up to 3 years
Incidence of cancer | up to 3 years
The change from baseline in vital signs and laboratory data | Baseline and 3 months, 6 months, 1 year, 2 years, 3 years after administration
Incidence of other adverse events | up to 3 years
Incidence of drug-related adverse events | up to 3 years
Incidence of serious adverse events | up to 3 years
The change from baseline in HbA1c | Baseline and 3 months, 6 months, 1 year, 2 years, 3 years after administration
The change from baseline in Fasting Plasma Glucose | Baseline and 3 months, 6 months, 1 year, 2 years, 3 years after administration